CLINICAL TRIAL: NCT03486821
Title: Pilot Trial of Ultra-hypofractionated Radiation in Early Prostate Cancer
Brief Title: Ultra-hypofractionated Radiation in Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Xinglei Shen, Medical Doctor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2017-PROS-UltraHypoFracRT
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Early Stage Prostate Cancer
Keywords: Radiation Therapy; ultra-short Radiation; SBRT; prostate; quality of life; financial toxicity
MeSH Terms: conditions — Financial Stress | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hypofrac Radiation Therapy (Experimental): All patients on this study will receive the same type of therapy, 2 treatment hypofractionated radiation therapy.
  Radiation treatment will start approximately 1-2 weeks after the simulation scan. Prior to each treatment, you will be asked to have a full bladder and empty rectum. You will be asked to take a liquid diet starting the afternoon prior to each treatment, and a laxative (such as Miralax) in the evening prior to each treatment. You will also be asked to take a Fleet's enema about 1 hours prior to the treatment time to ensure that the rectum is empty. To ensure full bladder, you will be asked to drink about 32 oz of water after the enema. This is the same procedure as above for the prep before the simulation scan.
  Each treatment should take about 10-20 minutes.
  Interventions: Radiation: Hypofractionated Radiation

INTERVENTIONS:
Radiation: Hypofractionated Radiation — All patients on this study will receive the same type of therapy, 2 treatment hypofractionated radiation therapy.

SUMMARY:
The primary objective of this study is to demonstrate that ultra-hypofractionation of prostate cancer does not increase urinary toxicity as defined by the EPIC-26 GU domain patient reported outcome.

DETAILED DESCRIPTION:
This is a pilot clinical trial looking at 2 fraction SBRT radiation therapy as an alternative to standard of care. Data does not yet exist for the safety and efficacy of this regimen.

However, the feasibility of ultra-short radiation therapy treatments has already been demonstrated in an analogous treatment using high-dose rate (HDR) brachytherapy. HDR brachytherapy has been adopted at high volume cancers centers as a standard treatment for prostate cancer. Typical doses have been 26 - 27 Gy over 2 fractions (13 or 13.5 Gy per fraction). Overall, toxicity and efficacy of HDR brachytherapy have compared favorably to other treatment modalities.

Dosimetric planning models between SBRT and HDR brachytherapy suggest minor differences. HDR brachytherapy was able to achieve higher intraprostatic maximum doses and lower rectal doses, but target volume coverage and urethral dose was not significantly different. These data suggest that reducing SBRT treatments from 5 fractions to 2 fractions may be feasible, efficacious and tolerable.

Eligible patients include all patients who are otherwise eligible for standard 5 fraction SBRT prostate. Study population will be low and intermediate patients with good urinary function (as defined by small prostate volume and low IPSS score). SBRT treatment will be delivered to the prostate to 12.5 Gy x 2 fractions.

Hormonal therapy is permitted on this study. Permitted agents include: leuprolide (Lupron/Eligard), biclutamide (Casodex), and degarelix (Firmagon).

Rectal sparing with hydrogel spacer (SpaceOAR) will be encouraged.

All patients will be enrolled with interim safety analyses after every occurrence of a grade 3 acute or late toxicity. Interval safety analysis will also be performed for recurrence and decrease in EPIC GU domain quality of life. Biospecimen and financial toxicity data will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant to sign a written informed consent.
* Diagnosed with prostate cancer, T1-T2bN0M0 GS6-7, PSA < 20
* IPSS score < 15 (and < 10 if on medication for benign prostatic hypertrophy such as tamsulosin) at time of enrollment (Appendix 21.4)
* Prostate volume (by US, CT or MRI measurement) < 50 cc at time of enrollment
* Androgen deprivation therapy based on clinician judgment is permitted on study
* Life expectancy > 10 years based on clinician's judgment
* No other active malignancy
* Age ≥ 18 years
* Performance Status Eastern Cooperative Oncology Group (ECOG) 0-1 (Appendix 21.5).
* Other study-specific criteria:
* Men of child-bearing potential must not donate sperm while on this study and for 90 days after their last study treatment.

NOTE: Acceptable forms of birth control are listed below:

* One Barrier method (cervical cap with spermicide plus male condom; diaphragm with spermicide plus male condom) PLUS
* Hormonal method (oral contraceptives, implants, or injections) or an intrauterine device (e.g., Copper-T).

Exclusion Criteria:

* Current or anticipated use of other investigational agents while participating in this study.
* Psychiatric illness/social situations that would limit compliance with study requirements
* Prior pelvic radiation therapy
* Prior prostatectomy
* Inflammatory bowel disease or connective tissue disease requiring medical management

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Toxicity Rates | up to 5 year post radiation
  Patient reported urinary function, as defined by the EPIC-26 GU domain patient reported outcome for prostate cancer patients

SECONDARY OUTCOMES:
Biochemical Control Rate | 1 month post-Radiation Therapy (RT), every 3 months- post RT for the first year and then every 6 months post RT for the next 4 years
  Biochemical freedom from progression as defined by ASTRO Phoenix criteria at 3 years
Radiation Therapy Oncology Group (RTOG) Late Toxicity Rate | 3 year
  Rate of Grade 3+ gastrointestinal (GI) or genitourinary (GU) late toxicity at 3 years as defined by RTOG late toxicity scored on a 1 to 4 scale with a higher value representing a worse outcome.
RTOG Acute Toxicity Rate | 90 days
  Rate of Grade 2+ GI or GU acute toxicity within 90 days of treatment as defined by RTOG acute toxicity scored on a 1 to 4 scale with a higher value representing a worse outcome.
Oxidative stress as a predictor of toxicity | 1 month post-RT, every 3 months- post RT for the first year and then every 6 months post RT for the next 4 years
  exploring the oxidative stress markers of the patient to use as a predictor of acute and late toxicty
Financial Toxicity Measurement | 3 months, 6 months, and 12 month visits only
  Determined by evaluation of patient completion of questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Xinglei Shen, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center/ Cancer Center, Kansas City, Kansas, United States